CLINICAL TRIAL: NCT01957605
Title: Study of Hemodynamic Variations During Prone Position Surgery: Measurement of Mean Systemic Pressure and Venous Return Resistance
Brief Title: Mean Systemic Pressure Measurement During Prone Position Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5673
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Hemodynamic Variation During Surgery
Keywords: prone position; hemodynamic variation; mean systemic pressure

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prone position: Patient scheduled for surgery in the prone position

SUMMARY:
Venous return is driven by the pressure gradient between mean systemic pressure and right atrial pressure. However, mean systemic pressure is more a physiological concept than an available clinical measurement. Indeed, the mean systemic pressure is the one that would be measured anywhere within the vascular system after cardiac arrest. Recent advances in hemodynamic monitoring have made MSP available to the clinician through beat-by-beat cardiac output measurements during respiratory pauses under mechanical ventilation. In this way, it is possible to calculate MSP, the pressure gradient and the venous return resistances. The investigators aim is to explain the hemodynamic variations and the decrease in cardiac output observed during prone position. The investigators hypothesis is that venous return resistances are increased during prone position probably following an increased intra-abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Prone position neurosurgery
* High-risk neurosurgery

Exclusion Criteria:

* Emergency surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for neurosurgery in the prone position
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
mean systemic pressure variation | during surgery after the patient is put in prone position
  change of mean systemic pressure from supine position to prone position during surgery

SECONDARY OUTCOMES:
intrathoracic pressure variation | during surgery during surgery after the patient is put in prone position
  Change of intrathoracic pressure from supine position to prone position during surgery
intravesical pressure variation | during surgery during surgery after the patient is put in prone position
  Change of intravesical pressure from supine position to prone position during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Julien Pottecher, MD, Principal Investigator — University Hospital of Strasbourg
Locations (1):
- University Hospital of Strasbourg, Strasbourg, France